CLINICAL TRIAL: NCT02240940
Title: PARACHUTE China: Multi-center, Prospective, Single-arm Clinical Evaluation of the Safety and Efficacy of the Parachute Percutaneous Left Ventricle Partitioning System
Brief Title: PARACHUTE China Approval Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company closed
Sponsor: CardioKinetix, Inc (Industry)
Collaborators: Guangzhou Chuangsi Medical Technology Co., Ltd. (Unknown); Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD1735
Record Dates: First submitted 2014-09-05; First posted 2014-09-16 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Heart Failure
Keywords: Heart Failure; Volume Reduction; Pressure Reduction; Ischemic Heart Failure; LAD Infarct
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Parachute Implant (Experimental): Appropriate patients meeting inclusion / exclusion will be implanted with the Parachute device after screening with transthoracic echocardiography (TTE) and cardiac CT or MRI.
  Interventions: Device: Parachute Implant

INTERVENTIONS:
Device: Parachute Implant — CardioKinetix's Parachute implant device is suitable for use in isolating the dysfunctional region of the left ventricle in patients with symptoms of heart failure due to ischemic heart disease. Potential benefits of the Parachute implant device are improvement in hemodynamics and the clinical symptoms of heart failure.

SUMMARY:
The design of this study is a multi-center, prospective, single-arm clinical trial to evaluate the safety and efficacy of the Parachute percutaneous left ventricle partitioning system. The purpose of this trial is to use the Parachute percutaneous left ventricular partitioning system to isolate the malfunctioning portion of the left ventricle in patients with symptoms of heart failure due to ischemic heart disease and provide the data required to gain Chinese regulatory approval.

DETAILED DESCRIPTION:
CardioKinetix has developed a catheter-based treatment method that can be used for treating patients with heart failure due to ischemic heart disease (left ventricle enlargement after anterior wall myocardial infarction). This implant device, called the "Parachute," is a partitioning membrane placed inside the apex of an enlarged ventricle with motion abnormalities. The Parachute implant device can then isolate the dysfunctional apex region in the ventricle, reduce ventricular volume, and improve left ventricular diastolic compliance.

Patients approved for enrollment after screening by cardiac CT or MRI will be implanted with a Parachute implant device (the study device). Patients will receive all appropriate medical therapy (AAMT) approved by their physician.

The patient cohort will include patients with heart failure who have wall motion abnormalities due to previous myocardial infarction, left ventricular ejection fraction ≤40% and ≥15%, and NYHA class II - IV（non-hospitalized). A maximum of 30 patients will be enrolled at seven centers. Patients who have passed screening with transthoracic echocardiography (TTE) and cardiac CT or MRI will be enrolled in the trial.

After confirming that a patient meets the enrollment qualifications with cardiac CT or MRI evaluation, the patient will be enrolled in the trial and will be implanted with a Parachute device and treated with warfarin/aspirin anticoagulation therapy.

In the follow-up periods 3 months, 6 months, and 1 year after surgery, clinical evaluation, TTE testing, functional assessment, 6-minute walk test, and evaluation of adverse events will be done.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ≤ 79 years
* BMI < 40'
* Left ventricle ejection fraction ≤40% and ≥15%
* Previous transthoracic echocardiography showing LV MI structural heart dysfunction represented by LV wall motion abnormalities (WMA)
* Appearance of ischemic heart failure symptoms (NYHA class II to "nonhospitalized" class IV) following anterior wall infarction and within the previous 60 days
* Left ventricle must have the appropriate anatomical structures (size and shape); cardiac CT and left ventricular angiography are used to confirm that implanting an appropriate Parachute device is possible
* Have received appropriate treatment according to ACC/AHA guidelines
* Subject or his/her legal representative informed of the nature of the study and consented to participate in all the provisions of the trial, signed the EC-approved informed consent form, agreed to undergo the post-surgery treatment plan and follow-up requirements, and is able to complete the follow-up and required follow-up examinations.

Exclusion Criteria:

* Significant ventricle wall motion abnormalities in addition to the anteroapical region
* Valvular stenosis or regurgitation (tricuspid, aortic, or mitral valve) > 2+
* Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* Requires long-term dialysis for end-stage renal disease or onset of sepsis or active endocarditis
* Life expectancy at time of enrollment and hospitalization <1 year
* Known allergies or contraindications to aspirin, heparin, warfarin, nitinol (titanium and nickel alloy), or sensitivity to contrast agents, that cannot be sufficiently treated with medication before surgery
* Cardiogenic shock within 72 hours of screening
* Pregnant or planning to become pregnant during the study period
* Participated in a clinical trial of another drug or medical device within 30 days of screening
* The researchers have determined that patient compliance is poor and that the person will be unable to complete the study in accordance with the requirements

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Reduction of LVESVi | 3 months
  The primary outcome measure is comparison of reduction in left ventricle end systolic volume index（LVESVi) after 3 months with baseline LVESVi. Evaluation will be performed via transthoracic echocardiography (TTE) by an independent central ultrasound laboratory (Yale University Clinical Research).

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 3 months
  Major adverse cardiac events (MACE) are defined as death from any cause, myocardial infarction, need for elective or urgent cardiac or thoracic aortic surgery or need for use of device or device surgery with a catheter as the basis of interventional therapy, or total renal failure requiring dialysis. The Kaplan-Meier method will be used to evaluate event-free survival after Parachute implantation.
Improvement in NYHA Class | 3 months
  All patients will undergo NYHA class evaluation at each time point. At the 3-month follow-up visit, the percentage of patients who have improvement in NYHA class (an improvement of at least 1 in comparison with NYHA class at baseline) will be measured.
Improvement in 6 minute walk test | 3 months
  The difference in the distance of the 6-minute walk will be measured by comparing the distance walked at the 3-month follow-up visit with the baseline distance walked.
Improvement in Quality of Life | 3 months
  The difference in EQ5D score by comparing EQ5D score at the 3-month follow-up visit with the EQ5D score at baseline will be measured.
Procedural Success | Day 0
  Technical success: Success in releasing the Parachute implant or successful completion of surgery.
  Combined success：The release of all devices with no serious adverse events, additional intervention surgeries, embolisms, technical failures (displacement, loss, etc.) or other problems.

OTHER OUTCOMES:
Long-term Safety | 6 months and 1 year
  Patients will be invited to continue participating in an extended observation study at 6 and 12 months. Patients who agree to participate 6 months and 12 months after surgery will receive the same evaluations as described in the 3-month follow-up visit.
  Descriptive reports of safety will be made using all the information gathered through the core research and the additional information from the extended observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Study Chair — Chinese Academy of Medical Sciences, Fu Wai Hospital; Yuejin Yang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fu Wai Hospital; Yuong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (7):
- China (7):
  - Chinese Academy of Medical Sciences Fu Wai Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang
  - 10th People's Hospital Affiliated to Tongji University, Shanghai
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai
  - Zhongshang Hospital of Fudan University, Shanghai
  - General Hospital of Shenyang Military Region, Shenyang

REFERENCES:
- [Derived] Li J, Liu H, Liu Q, Liu C, Xiong W, Ma W, Zhang B, Dong S, Li T. Long-term prognosis analysis of PARACHUTE device implantation in patients with ischemic heart failure: a single-center experience of Chinese patients. J Cardiothorac Surg. 2021 Apr 20;16(1):98. doi: 10.1186/s13019-021-01484-0. PMID 33879206
- [Derived] Yang YJ, Huo Y, Xu YW, Wang JA, Han YL, Ge JB, Zhang RY, Yan XY, Gao RL. Percutaneous Ventricular Restoration Therapy Using the Parachute Device in Chinese Patients with Ischemic Heart Failure: Three-Month Primary End-point Results of PARACHUTE China Study. Chin Med J (Engl). 2016 Sep 5;129(17):2058-62. doi: 10.4103/0366-6999.189048. PMID 27569231